CLINICAL TRIAL: NCT06837792
Title: The Exploratory Randomized Phase II Study of Trastuzumab Deruxtecan Versus Endocrine Therapy of Physician's Choice in Low-HER2 Expressing Hormone Receptor-positive Advanced Breast Cancer Patients
Brief Title: Trastuzumab Deruxtecan vs Endocrine Therapy in Low-HER2 HR+ Advanced Breast Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2023-1363
Record Dates: First submitted 2024-06-12; First posted 2025-02-20 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Hormone Receptor(HR)-Positive, Low HER2 Advanced Breast Cancer Patients (HER2 IHC 1+ or 2+ & ISH Negative)
Keywords: low HER2, advanced breast cancer, T-DXd

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental treatment arm(T-DXd arm) (Experimental): Trastuzumab deruxtecan (T-DXd)
  Interventions: Drug: Experimental treatment arm
- Control treatment arm (Active Comparator): Endocrine therapy of physician's choice[TPC]
  Interventions: Drug: Control treatment arm

INTERVENTIONS:
Drug: Experimental treatment arm — Trastuzumab deruxtecan (T-DXd) 5.4mg/kg intravenous infusion every 3 weeks.
  (1 cycle = 3 weeks)
  Other Names: T-DXd arm
  Arms: Experimental treatment arm(T-DXd arm)
Drug: Control treatment arm — 1. Fulvestrant intramuscular injection of two 250mg injection every 4 weeks (every 2 weeks for the first cycle, 1 cycle = 4 weeks)
  2. Fulvestrant (administered same as above) + alpelisib 300mg oral administration every day
     (1 cycle = 4 weeks)*
  3. Exemestane 25mg oral administration every day (1 cycle = 4 weeks)
  4. Exemestane 25mg + everolimus 10mg oral administration every day (1 cycle = 4 weeks)
  5. Tamoxifen 20mg oral administration every day (1 cycle = 4 weeks)
  6. Fulvestrant (administered same as above) + Capivasertib 400mg oral administration twice a day(dosed on Days 1 to 4 in each week of a 28-day treatment cycle)
     * fulvestrant + alpelisib can be selected in PIK3CA activating mutation positive patients
     * Fulvestrant + Capivasertib can be selected in 1 or More mutation positive of PIK3CA/AKT1/PTEN
  Other Names: Endocrine therapy of physician's choice[TPC]
  Arms: Control treatment arm

SUMMARY:
"This is a randomized phase II, two-arm, open label, clinical trial to identify LP-WGS ctDNA biomarker to predict T-DXd response in low-HER2 expressing advanced breast cancer patients compared with endocrine therapy. The hormone receptor (HR)-positive low-HER2 advanced breast cancer patients (HER2 IHC 1+ or 2+ & ISH negative, n=141) who progressed on 1st line endocrine + CDK4/6 inhibitor therapy and received no other systemic therapy for advanced disease are enrolled in this study. Patients are 2:1 randomized to receive T-DXd (5.4mg/kg every 3 weeks, n=94) or endocrine therapy of physician's choice (TPC: fulvestrant, fulvestrant + alpelisib, Fulvestrant + Capivasertib, exemestane, exemestane + everolimus, or tamoxifen, n=47, fulvestrant + alpelisib can be selected in PIK3CA activating mutation positive patients, Fulvestrant + Capivasertib can be selected in 1 or More mutation positive of PIK3CA/AKT1/PTEN). The mandatory baseline archival tissue and ctDNA collection followed by on-treatment ctDNA collection (Cycle 1, Cycle 2, and Cycle 6) and ctDNA collection at progression will be performed in this study.

The primary endpoint is PFS after randomization in two treatment arms. The secondary endpoints include overall survival (OS), objective response rate (ORR), progression-free survival (PFS2), adverse events by CTCAE 5.0 criteria, and Quality of life (QoL) measured by EORTC-QLQ-C30 and EORTC-QLQ-BR23 evaluated by questionnaire. The exploratory endpoints are to identify ctDNA biomarkers to predict the TDxd treatment outcome (PFS, OS, ORR) compared to endocrine therapy in HER2-low advanced breast cancer patients and to assess the accordance of genomic profiles between ctDNA and tumor tissues. Predictive biomarkers include copy number aberration (CNA) of gene loci, total ctDNA CNA burden, mutations, ctDNA-based molecular subtype, or HER2 amplicon copy number on LP-WGS ctDNA analysis. The investigator believe this trial will identify crucial circulating biomarkers for T-DXd treatment response in low-HER2 patients, which can guide right patient selection and potential molecular target identification to maximize T-DXd response and to overcome T-DXd resistance.

DETAILED DESCRIPTION:
Study Design: Randomized phase II, two-arm, randomized, open label study

- The Hormone receptor (HR)-positive HER2-low advanced breast cancer patients (HER2 IHC 1+ or 2+ & ISH negative, n=141) who progressed on first-line endocrine + CDK4/6 inhibitor therapy for advanced disease will be enrolled in this study. Patients will be 2:1 randomized to experimental and control treatment arms by stratification factors below

Stratification factor

1. Visceral metastasis (with visceral metastasis versus without visceral metastasis)
2. Progression-free survival on prior CDK4/6 inhibitor therapy (< 6 months versus ≥ 6 months)

   * In the experimental treatment arm (n=94), patients receive trastuzumab deruxtecan (T-Ddx) 5.4mg/kg intravenous infusion every 3 weeks. In the control treatment arm (n=47), patients receive endocrine therapy of physicians' choice (TPC: fulvestrant, fulvestrant + alpelisib, exemestane, exemestane + everolimus, or tamoxifen; fulvestrant + alpelisib can be selected in PIK3CA activating mutation positive patients). The study treatment will continue until disease progression by RECIST 1.1, unacceptable toxicity, end of study, or death.
   * This study both enrolls pre- and post-menopausal patients, and pre-menopausal patients should receive ovarian function suppression treatment (GnRH agonist injection or surgical bilateral oophorectomy) while receiving fulvestrant or aromatase inhibitor treatment in the control arm.
   * The endocrine TPC is pre-selected by investigator in screening period before randomization. The regimens that the patient received for advanced disease before cannot be selected. The regimen that the patients received for (neo)adjuvant therapy for breast cancer before cannot be selected unless the recurrence of disease was diagnosed > 1 year after the completion of the (neo)adjuvant therapy.
   * The evaluation of tumor response by computed tomography or magnetic resonance imaging of the chest, abdomen, and pelvis will be performed every 9 weeks from the date of randomization for 54 weeks and performed every 12 weeks after then until objective (RECIST 1.1 defined) disease progression.
   * Mandatory baseline tissue and ctDNA collection followed by three on-treatment ctDNA samples (Day 1 of Cycle 2, Cycle 3, and Cycle 6) will be collected. The post-treatment ctDNA (mandatory) and tumor tissues (optional) will be also collected
   * The patient samples will be evaluated to identify predictive biomarkers including copy number aberration (CNA), mutations, molecular subtype, or HRD status on LP-WGS ctDNA analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed hormone receptor-positive advanced breast cancer patients

   1. Have recurrent, metastatic, or unresectable disease
   2. Have HER2-low expression status, defined as IHC 2+/ISH- or IHC 1+,with a validated assay by ASCO/CAP guidelines
   3. Have no previous history of HER2-positive breast cancer (IHC 3+ or ISH+) by ASCO/CAP guidelines
   4. The hormone receptor (HR) status is defined by ER/PR IHC nuclear staining, and ER or PgR ≥1% is defined as hormone receptor-positive status
2. Patients who progressed on 1st line endocrine + CDK4/6 inhibitor therapy for advanced breast cancer and received no other systemic therapy for advanced breast cancer. The all FDA-approved CDK4/6 inhibitors (palbociclib, ribociclib, and Abemaciclib) are allowed, and combination with aromatase inhibitors or fulvestrant are both allowed.
3. Patients who have received chemotherapy or adjuvant endocrine therapy in the neo-adjuvant or adjuvant setting are eligible.
4. Female patients with ≥19 years of age
5. Radiologic or objective evidence of disease progression on or after the last systemic therapy prior to starting study treatment
6. Patients must have at least one measurable lesion by RECIST 1.1 criteria, which was not previously irradiated or showed objective progression after irradiation to that lesion
7. Patients must have an adequate tumor tissue sample available for assessment of HER2 by central laboratory and other exploratory biomarker analyses
8. Patients with ECOG performance status 0 or 1
9. Both pre- and post-menopausal patients are eligible, and pre-menopausal patients should receive ovarian function suppression treatment (GnRH agonist injection or surgical bilateral oophorectomy) while receiving fulvestrant or aromatase inhibitor treatment in the control arm.
10. Adequate organ function for treatment Adequate organ and bone marrow function within 14 days before randomization/enrolment as described below:"

    a) Haemoglobin: ≥ 9.0 g/dL NOTE: Participants requiring ongoing transfusions or growth factor support to maintain haemoglobin ≥9.0 g/dL are not eligible. (Red blood cell transfusion is not allowed within 1 week prior to C1D1) b) Serum albumin: ≥ 2.5 g/dL c) International normalised ratio or Prothrombin time and either partial thromboplastin or activated partial thromboplastin time: ≤ 1.5 × ULN d) Absolute neutrophil count (ANC) ≥1500 cells/mm3
    * granulocyte-colony stimulating factor administration is not allowed within 1 week prior to C1D1 ) e) Platelets ≥100,000 cells/mm3
    * Platelet transfusion is not allowed within 1 week prior to C1D1) f) Estimated creatinine clearance ≥50 mL/min, or serum creatinine <1.5x institution upper limit of normal (ULN) g) Bilirubin≤1.5 x ULN
    * if no liver metastases or < 3×ULN in the presence of documented Gilbert's syndrome (unconjugated hyperbilirubinemia) or liver metastases at baseline h) AST (SGOT) ≤2.5 x ULN (5.0 x ULN if hepatic metastases) i) ALT (SGPT) ≤2.5 x ULN (5.0 x ULN if hepatic metastases)
11. 12-Lead electrocardiogram (ECG) with normal tracing or non-clinically significant changes that do not require medical intervention
12. QTc interval ≤470 msec and without history of Torsades de pointes based on average of the screening triplicate 12-lead ECG
13. Pointes or other symptomatic QTc abnormality
14. LVEF (by MUGA or echocardiogram) of ≥50% within 28 days before randomization/enrollment
15. No history of pneumonitis other than radiation pneumonitis
16. The patient has provided signed informed consent
17. Neither pregnant or breastfeeding female patients
18. Fertile women who are not in pregnancy or breastfeeding should use effective contraception for a period from two weeks before the start of research treatment, during treatment and up to seven months after last dose of study treatment
19. No other concurrent severe and/or uncontrolled medical disease which could compromise study participation, including any of the following:
20. Adequate treatment washout period before enrollment are below -Major surgery ≥ 4 weeks -Radiation Therapy including palliative stereotactic radiation therapy to chest ≥ 4 weeks -Palliative stereotactic radiation therapy to other anatomic areas including whole brain radiation ≥ 2 weeks -Anti-Cancer chemotherapy [Immunotherapy (non-antibody based therapy)], retinoid therapy, hormonal therapy ≥ 3 weeks -Antibody based anti-cancer therapy ≥ 4 weeks -Targeted agents and small molecules ≥ 2 weeks or 5 half-lives, whichever is longer -Nitrosoureas or mitomycin C ≥ 6 weeks -Chloroquine/Hydroxychloroquine ≥ 14 days -Cell-free and CART, peritoneal shunt or drainage of pleural effusion, ascites or pericardial effusion ≥ 2 weeks prior to screening assessment

Exclusion Criteria:

1. Previous history of T-DXd or Dato-Dxd treatment for advanced breast cancer
2. Severe Cardiac disease (e.g., uncontrolled hypertension, congestive cardiac failure, ventricular arrhythmias, active ischemic heart disease, myocardial infarction within the past year, Left Ventricular Ejection Fraction (LVEF) > grade 2)
3. Patients with a medical history of myocardial infarction (MI) within 6 months before randomization/enrolment, symptomatic congestive heart failure (CHF) (New York Heart Association Class II to IV), Subjects with troponin levels above ULN at screening (as defined by the manufacturer), and without any myocardial related symptoms, should have a cardiologic consultation before enrollment to rule out MI.
4. Current active hepatic or biliary disease (except for Gilbert syndrome, asymptomatic gallstones, liver metastasis or stable chronic liver disease per investigator assessment)
5. Uncontrolled infection requiring IV antibiotics, antivirals, or antifungals
6. Receipt of live, attenuated vaccine (mRNA and replication deficient adenoviral vaccines are not considered attenuated live vaccines) within 30 days prior to the first dose of T-DXd.
7. Has unresolved toxicities from previous anticancer therapy, defined as toxicities (other than alopecia) not yet resolved to Grade ≤ 1 or baseline.

   Note: Subjects may be enrolled with chronic, stable Grade 2 toxicities (defined as no worsening to >Grade 2 for at least 3 months prior to [randomization/enrollment/Cycle 1 Day 1] and managed with standard of care treatment) that the investigator deems related to previous anticancer therapy, such as:
   * Chemotherapy-induced neuropathy
   * Fatigue
   * Residual toxicities from prior IO treatment: Grade 1 or Grade 2 endocrinopathies which may include:

     1. Hypothyroidism/hyperthyroidism
     2. Type 1 diabetes
     3. Hyperglycaemia
     4. Adrenal insufficiency
     5. Adrenalitis
     6. Skin hypopigmentation (vitiligo)
8. Lung-specific intercurrent clinically significant illnesses including, but not limited to, any underlying pulmonary disorder (i.e., pulmonary emboli within three months prior to study enrollment, severe asthma, severe chronic obstructive pulmonary disorder [COPD], restrictive lung disease, significant pleural effusion etc.), and any autoimmune, connective tissue or inflammatory disorders with pulmonary involvement (i.e.,rheumatoid arthritis, Sjogren's syndrome, sarcoidosis etc.), and/or prior pneumonectomy.
9. Has as a history of (non-infectious) ILD/ pneumonitis, has current ILD/pneumonitis, or where suspected ILD/pneumonitis cannot be ruled out by imaging at screening.Presence of spinal cord compression, symptomatic CNS metastases, or CNS metastases that require local CNS-directed therapy (such as radiotherapy or surgery). Patients with treated brain metastases should be neurologically stable (for 4 weeks post treatment and prior to study enrollment) and without steroid therapy over physiologic dose (> 10mg prednisolone/day) for at least 2 weeks before administration of study drug.
10. Significantly altered mental status prohibiting the understanding of the study, or with psychological, familial, sociological, or geographical condition potentially hampering compliance with the study protocol and follow-up schedule
11. Active primary immunodeficiency, known human immunodeficiency virus (HIV) infection, or active hepatitis B or C infection. Subjects with past or resolved hepatitis B virus (HBV) infection who are anti-HBc positive (+) are eligible only if they are HBsAg negative (-). Patients positive for hepatitis C antibody are eligible only if polymerase chain reaction is negative for HCV RNA. Subjects should be tested for HIV prior to randomization/enrollment if required by local regulations or institutional review board (IRB)/ethics committee (EC).
12. Multiple primary malignancies within 5 years, except adequately resected non-melanoma skin cancer, curatively treated in-situ disease, other solid tumors curatively treated, or contralateral breast cancer.
13. Patients unable to swallow orally administered medication and patients with gastrointestinal disorders likely to interfere with absorption of the study medication.
14. Pregnant or breast-feeding women.
15. Previous allogeneic bone marrow transplant.
16. Patients with a known hypersensitivity to T-DXd
17. History of severe hypersensitivity reactions to other monoclonal antibodies
18. Prior treatment with antibody drug conjugate that comprised an exatecan derivative that is a topoisomerase I inhibitor

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female patients
Enrollment: 141 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
PFS according to RECIST 1.1 in the ITT population. | from date of randomization until the date of first evidence of disease progression or date of death from any cause, whichever came first, assessed up to 36 months
  Progression-free survival (PFS) is defined as the time from day 1 of the randomization to the first evidence of disease progression or death, whichever is earlier.

SECONDARY OUTCOMES:
OS | On treatment: Every 3-4 weeks from date of randomization until the date of of death from any cause, assessed up to 36 months
  OS measured from the time of randomization to the time of death of any cause.
ORR | From screening and every 9 weeks for 54 weeks from randomization and every 12 weeks after 54 weeks from randomization to objective (RECIST 1.1 defined) disease progression, withdrawal of subject consent, or unacceptable toxicity, up to 36 months
  Objective response rate as defined as the proportion of patients with at least 1 visit response of partial response or complete response based on RECIST 1.1 by investigator assessment
Progression-free survival (PFS2) | from date of randomization until the date of first evidence of second disease progression or date of death from any cause, whichever came first, assessed up to 36 months
  PFS2 as defined time from randomization until second progression on next-line of treatment, as assessed by investigator or death due to any cause
safety | From administration of the first dose of study treatment and every 3-4 weeks on treatment and until 90 days after the last administration of the investigational drug or the initiation of new antitumor therapy, up to 36 months
  Adverse events by CTCAE 5.0 criteria.
Quality of life (QoL) by EORTC-QLQ-C30 | From administration of the first dose of study treatment and every 9 weeks (±3 days) until 2 years (even after disease progression))
  Quality of life (QoL) measured by EORTC-QLQ-C30 evaluated by questionnaire
Quality of life (QoL) by ORTC-QLQ-BR23 | From administration of the first dose of study treatment and every 9 weeks (±3 days) until 2 years (even after disease progression))
  Quality of life (QoL) measured by EORTC-QLQ-BR23 evaluated by questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Medical Oncology, Yonsei Cancer Center, Yonsei Univ. College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No